CLINICAL TRIAL: NCT07318961
Title: Visual and Anatomical Outcomes of Autologous Tenon's Capsule Graft for Refractory Macular Holes
Brief Title: Autologous Tenon's Capsule Graft for Refractory Macular Holes
Acronym: ATCG-RMH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ehab Mohamed Elsayed Mohamed Saad, Lecturer, Benha University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Macular hole rapair
Record Dates: First submitted 2025-12-21; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Macular Hole Surgery
Keywords: Autologous Tenon's Capsule Graft; Macular Hole
MeSH Terms: conditions — Retinal Perforations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autologous Tenon's Capsule Graft (Other): Procedure
  Interventions: Procedure: Autologous Tenon's Capsule Graft Placement

INTERVENTIONS:
Procedure: Autologous Tenon's Capsule Graft Placement — Participants will undergo 23-gauge pars plana vitrectomy. Autologous Tenon's capsule tissue will be harvested through conjunctival peritomy, trimmed appropriately, and placed into the macular hole using intraocular forceps. Perfluorocarbon liquid may be used for graft stabilization, followed by silicone oil tamponade. Silicone oil removal is planned after 8-12 weeks.

SUMMARY:
This prospective interventional study evaluates the anatomical and functional outcomes of autologous Tenon's capsule grafting in patients with refractory full-thickness macular holes. Eligible patients include those with chronic large macular holes (>400 µm) or persistent holes following prior pars plana vitrectomy with internal limiting membrane peeling and gas tamponade. Anatomical closure will be assessed using spectral-domain optical coherence tomography, and functional outcomes will be evaluated by best-corrected visual acuity over a 3-month follow-up period.

DETAILED DESCRIPTION:
Refractory full-thickness macular holes represent a significant surgical challenge, with reduced closure rates following conventional techniques, particularly in large or chronic defects. Autologous tissue grafting has emerged as an alternative strategy to provide a biological scaffold for retinal tissue bridging and gliosis. Tenon's capsule is a readily accessible autologous fibrovascular tissue that can be harvested intraoperatively with minimal morbidity.

This prospective single-arm clinical study aims to assess the anatomical closure rate and visual outcomes following autologous Tenon's capsule graft placement in refractory macular holes. All patients will undergo standard pars plana vitrectomy, placement of a trimmed Tenon's graft into the macular hole, and silicone oil tamponade. Outcomes will be evaluated using standardized visual acuity testing and spectral-domain OCT imaging at predefined postoperative intervals.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Refractory full-thickness macular hole defined as:
* Chronic macular hole >400 µm, or
* Persistent macular hole following prior vitrectomy with ILM peeling and gas tamponade
* Clear ocular media and adequate fixation for OCT imaging
* Ability to provide informed consent

Exclusion Criteria:

* Active ocular infection or inflammation
* Advanced glaucoma or optic neuropathy
* History of intraocular tumors
* Severe proliferative vitreoretinopathy
* Significant systemic diseases likely to affect visual recovery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-14 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-03 (Estimated)

PRIMARY OUTCOMES:
Macular hole anatomical closure | 3 months postoperatively
  Complete closure of the macular hole as confirmed by spectral-domain OCT

SECONDARY OUTCOMES:
Change in Best-Corrected Visual Acuity (logMAR) | Baseline (preoperative), 1 month postoperatively, and 3 months postoperatively
  Change in best-corrected visual acuity (BCVA), measured in logMAR units, comparing postoperative values with baseline (preoperative) BCVA to assess functional visual improvement following autologous Tenon's capsule graft surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Benha University, Banhā, Benha, Egypt